CLINICAL TRIAL: NCT03794375
Title: Impact of Primary Care Transfer for Thyroid Cancer Patients
Brief Title: Primary Care Transfer for Thyroid Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 95392418300005327
Record Dates: First submitted 2018-12-28; First posted 2019-01-07 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Differentiated Thyroid Cancer
Keywords: Follow-up; Telehealth; Recurrence
MeSH Terms: conditions — Recurrence | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (Active Comparator): The patients will remain in care at the HCPA thyroid disease outpatient clinic during the study period. This follow-up will be done by endocrinologists, and the patients will undergo clinical, biochemical (TSH, thyroglobulin, and antithyroglobulin) and radiological (cervical ultrasound) tests to seek disease recurrence. The patient's consultation will be done one or twice a year.
  Interventions: Other: Usual care
- Telehealth (Experimental): The patients will be discharged from the HCPA thyroid disease outpatient clinic, being instructed to seek the primary care level according to their place of residence to schedule a routine consultation in up to six months.
  After 45 days after the estimated date of the consultation (6 months after discharge), the Telehealth staff will contact the patient to check if the consultation was actually performed. When individuals report difficulty accessing the unit, contact will be made to the primary care teams and the Telehealth staff will schedule the appointment. A new contact will be made in 12 months to verify if the consultation was actually performed.
  Interventions: Other: Telehealth

INTERVENTIONS:
Other: Telehealth — After 45 days after the estimated date of the consultation (6 months after discharge), the Telehealth staff will contact the patient to check if the consultation was actually performed. When individuals report difficulty accessing the unit, contact will be made to the primary care teams and the Telehealth staff will schedule the appointment. A new contact will be made in 12 months to verify if the consultation was actually performed.
  Arms: Telehealth
Other: Usual care — The patients will remain in care at the HCPA thyroid disease outpatient clinic during the study period. This follow-up will be done by endocrinologists, and the patients will undergo clinical, biochemical (TSH, thyroglobulin, and antithyroglobulin) and radiological (cervical ultrasound) tests to seek disease recurrence. The patient's consultation will be done one or twice a year.
  Arms: Usual care

SUMMARY:
Introduction: Differentiated thyroid cancer (DTC) is the most common endocrine malignancy. It presents low recurrence rates (2-5%) and the consensus of DTC recommends long-term follow-up, without a definition of maximum follow-up time. The use of Telehealth is a strategy that aims to optimize the transition of care for patients from tertiary care to primary health care, helping to follow up these patients.

Objective: To evaluate the impact of the care transition between specialized care and primary health care of patients with DTC using telemedicine solutions.

Design / Patients: Randomized clinical trial. Patients with DTC with excellent response (without evidence of disease) after initial treatment.

Interventions / Outcomes: Patients will be randomized to follow-up in face-to-face consultations in tertiary care or transfer of care to primary care with support from the Telehealth Center of Rio Grande do Sul. After 18 months, all patients will be evaluated, the primary outcome being DTC recurrence rate. Outcomes related to quality of life and use of the health system will also be evaluated. Both follow-up strategies are expected to be equivalent, making it possible to optimize the use of the health system.

DETAILED DESCRIPTION:
Differentiated thyroid cancer (DTC) is the most frequent malignant neoplasm of the endocrine system, accounting for approximately 95% of the cases of carcinomas in this system. DTC is considered to be an indolent behavioral neoplasm with low rates of morbidity and mortality (mean survival in 10 years from 93 to 98%), being one of the malignancies with a greater chance of cure.

In recent years, the use of the initial treatment response, called "dynamic risk classification", has been advocated in order to better estimate the risk of unfavorable outcomes in patients with DTC. Using this classification, the recurrence rate in the contemporary CDT cohorts has been shown to be very low, at a household of 1-5%. In a cohort of our center, which evaluated 786 patients, the recurrence rate in the group of 357 patients classified as excellent response after the initial treatment was 2.8%, and none of these patients presented structural relapse (median follow-up of 4 years). Thus, it is possible to affirm that most of the patients classified as having an excellent response after initial treatment are permanently free of disease. However, the main consensus on the management of DTC recommends long-term follow-up, not defining the maximum follow-up time. This follow-up consists of consultations in specialized centers (preferably with endocrinologists), laboratory tests (TSH, thyroglobulin and antithyroglobulin antibody) and imaging.

In Brazil, the health network is characterized by the heterogeneity of hospital structures regarding the incorporation of technologies and service complexity, with a concentration of financial resources and specialized personnel in large cities and regional imbalance. Within this context, specialized outpatients with high complexity face overcrowding (of patients already under follow-up) and restricted access (to patients in need of follow-up). In this sense, transferring the care of follow-up patients in specialized hospitals to primary care level in their place of origin to maintain follow-up brings benefits to individuals and the system as a whole. The structure of referral of patients to the different levels of care in the Brazilian public health system occurs through the reference and counter-referral system, a fundamental point to guarantee the accessibility, universality, and integrality of care. It is understood as a counter-referral to a primary care level, with a lower degree of complexity, and should be the health unit closest to the patient's home. Facilitating mechanisms of reference and counter-reference processes are fundamental to guarantee the principle of integrality, adequate patient care and rational use of resources.

One of the formats for developing health care support and continuing education activities are teleconsulting, which are consultations recorded and performed among workers, health professionals and managers, through telecommunication instruments, with the purpose of clarifying doubts about clinical procedures, health actions and issues related to the work process. It is known that this type of systematic intervention based on practice is one of the most effective ways to promote permanent health education. The use of telehealth, through teleconsulting, for cases referred by primary care physicians to tertiary services is a strategy that aims to qualify and reduce referral lists for other medical professionals. Likewise, the use of telehealth emerges as a counter-referral strategy for patients already served by tertiary care for primary care units, ensuring patient and physician security of adequate management and assisted return for tertiary care, when necessary.

In this study, 206 patients with a diagnosis of DTC consecutively attended at the thyroid clinic of the Hospital de Clínicas of Porto Alegre and who presented excellent response to the initial treatment will be invited to participate in the study, and then randomized to two follow-up strategies:

1. Control group: patients will remain in care at the HCPA thyroid disease outpatient clinic;
2. Intervention group: outpatient discharge with telehealth support.

Patients with definitive postoperative hypoparathyroidism and/or postoperative vocal cord paralysis requiring tracheostomy will be excluded. All patients will be evaluated by the study team after completing 18 of follow-up. Clinical, laboratory (TSH, thyroglobulin and antithyroglobulin antibody) and imaging (cervical ultrasonography) for DTC relapse will be evaluated in this follow-up visit. The primary endpoint will be the DTC recurrence rate. This will be divided into biochemistry (when there are only signs of disease in laboratory tests) and structural (when demonstrated by clinical or imaging examination). Outcomes related to quality of life and use of the health system will also be evaluated. Both follow-up strategies are expected to be equivalent in relation to DTC recurrences, potentially enabling optimization of the use of the health system.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnostic of differentiated thyroid cancer and an excellent response to the initial treatment.

Exclusion Criteria:

* Definitive postoperative hypoparathyroidism.
* Postoperative vocal cord paralysis requiring tracheostomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 18 months
  All patients will be evaluated by the study team after completing 18 months of follow-up for this outcome. The presence of recurrence may be identified as a structural disease (evaluated by clinical examination and cervical ultrasound) or biochemical (evaluated by laboratory tests -thyroglobulin and antithyroglobulin antibody levels measurement). Both types of recurrence will be classified as an outcome.

SECONDARY OUTCOMES:
Patient's satisfaction evaluated by analogue-visual scale from 0 to 10. | 18 months
  This outcome will be evaluated by analogue-visual scale from 0 to 10.
Health care system access evaluated by the number of procedures related to the DTC performed by the patient. | 18 months
  This outcome will be evaluated by the number of procedures related to the DTC performed by the patient.
Hypothyroidism control evaluated by the TSH level during the follow-up of the patients. | 18 months
  This outcome will be evaluated by the TSH level during the follow-up of the patients.
Quality of life evaluated by EuroQol-5D (EQ-5D) | 18 months
  This outcome will be evaluated by EuroQol-5D (EQ-5D). The EuroQol-5D (EQ-5D) is a questionnaire that measures health status in five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. It is used to assess quality of life and can be used in a variety of health care applications.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael S. Scheffel, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Brazil

IPD SHARING:
Plan to Share IPD: Undecided